CLINICAL TRIAL: NCT02544204
Title: A Phase 2B Randomized Double Blind Placebo Controlled Study to Evaluate the Safety and Efficacy of JVS-100 Administered by Direct Intramuscular Injection as Adjunct to Revascularization of Infrapopliteal Lesions in Subjects With Advanced Peripheral Artery Disease and Tissue Loss
Brief Title: SDF1 Plasmid Treatment for Patients With Peripheral Artery Disease
Acronym: STOP-PAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juventas Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JTCS-007
Record Dates: First submitted 2015-08-06; First posted 2015-09-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 8 mg JVS-100 (Active Comparator): Biological/Vaccine: JVS-100 Injection Intramuscular Injection
  Interventions: Biological: JVS-100
- 8 mg placebo (Placebo Comparator): Biological/Vaccine: Placebo Injection Intramuscular Injection
  Interventions: Biological: Placebo
- 16 mg JVS-100 (Active Comparator): Biological/Vaccine: JVS-100 Injection Intramuscular Injection
  Interventions: Biological: JVS-100
- 16 mg placebo (Placebo Comparator): Biological/Vaccine: Placebo Injection Intramuscular Injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: JVS-100 — Biological/Vaccine: JVS-100 Intramuscular Injection
  Arms: 16 mg JVS-100; 8 mg JVS-100
Biological: Placebo — Biological/Vaccine: Placebo Intramuscular Injection
  Arms: 16 mg placebo; 8 mg placebo

SUMMARY:
To investigate the efficacy of the administration of JVS-100 delivered via direct intramuscular injections on a 3 month and 6 month composite endpoint of wound progression, healing and limb loss in patients with severe peripheral arterial disease with non-healing chronic wounds who undergo an open bypass grafting or endovascular procedure for treatment of infrapopliteal disease and are dosed within 12 days and 3 months following the procedure.

ELIGIBILITY:
Major Inclusion Criteria:

* Age ≥18
* Currently receiving standard of care wound treatment (>2 weeks) for chronic wounds or gangrene including as indicated: debridement, pressure offloading, infection control, and/or maintenance of a moist wound environment.
* Diagnosis of advanced PAD with tissue loss (ulceration and/or dry gangrene) on the foot of the index leg with an ulcer size of at least 0.5 cm2 and <25 cm2. Index wounds on the heel must be <10 cm2 that cannot be probed to bone, have exposed bone or osteomyelitis.
* Post revascularization intervention inclusion criteria include an attempt at open bypass grafting or endovascular intervention of a popliteal/infrapopliteal lesion(s) on the same leg that has tissue loss without significant improvement in TBI post intervention. The following will be accepted as demonstrating a lack of post intervention toe brachial index (TBI) improvement:

  * TBI ≤ 0.51or;
  * Toe pressure ≤50 mmHg with flat or dampened wave forms or;
  * Skin Perfusion pressure ≤40 mmHg at mid foot level or;
  * TcPO2 ≤40 mmHg
* Subjects willing to forgo treatment with hyperbaric oxygen, nerve stimulation or sympathectomy for the treatment of advanced PAD from time of consent to 6 months following the initial injection of study drug

Major Exclusion Criteria:

* Previous major amputation of the leg to be treated or planned major amputation or transmetatarsal amputation within the first month following enrollment.
* Only a short segment superficial femoral artery lesion - consistent with Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II) A or B category, and no infrapopliteal disease
* Staged or planned intervention in the index leg within 30 days after the index procedure
* Acute limb-threatening ischemia, trauma, known non-atherosclerotic vascular disease
* Non-salvageable limb defined as major tissue loss and an unsalvageable foot;
* Wounds that have decreased in size by >50% between the Screening visit and Day 0.
* If patient has active infection of the index limb that is being treated, and, in the opinion of treating physician, will not lead to an amputation within the next 3 months, the patient can be enrolled.
* Inability to safely perform a revascularization procedure due to uncontrolled diabetes or other medical condition.
* Presence of any other condition that, in the opinion of the investigator, might compromise any aspect of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The composite is designed to quantify clinically significant improvement or worsening over baseline by assigning a score to each patient that represents their overall outcome. | 3 months
  Change from baseline in the composite endpoint at 3 months in all treated (or one JVS-100 dose group) compared to all placebo.
The composite is designed to quantify clinically significant improvement or worsening over baseline by assigning a score to each patient that represents their overall outcome. | 6 months
  Change from baseline in the composite endpoint at 6 months in all treated (or one JVS-100 dose group) compared to all placebo.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Cardiovascular Associates of the Southeast, Birmingham, Alabama
  - UC Davis, Davis, California
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - MedStar Georgetown UH, Washington D.C., District of Columbia
  - Morton Plant Hosptial - Baycare, Clearwater, Florida
  - Mount Sinai Medical Center, Miami, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Northwestern, Chicago, Illinois
  - RUMC, Chicago, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Mayo, Rochester, Minnesota
  - Cardiology Associates Research, Tupelo, Mississippi
  - St. Luke's Mid America Heart Institute, Kansas City, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - UNC, Chapel Hill, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Summa Health, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Metro Health, Cleveland, Ohio
  - University Hospitals, Cleveland, Ohio
  - Lifespan Health System, Providence, Rhode Island
  - VCU, Richmond, Virginia
  - Medical College of Wisconsin, Milwauke, Wisconsin

REFERENCES:
- [Derived] Hammad TA, Rundback J, Bunte M, Miller L, Patel PD, Sadanandan S, Fitzgerald M, Pastore J, Kashyap V, Henry TD, Shishehbor MH. Stromal Cell-Derived Factor-1 Plasmid Treatment for Patients With Peripheral Artery Disease (STOP-PAD) Trial: Six-Month Results. J Endovasc Ther. 2020 Aug;27(4):669-675. doi: 10.1177/1526602820919951. Epub 2020 May 18. PMID 32419594
- [Derived] Shishehbor MH, Rundback J, Bunte M, Hammad TA, Miller L, Patel PD, Sadanandan S, Fitzgerald M, Pastore J, Kashyap V, Henry TD. SDF-1 plasmid treatment for patients with peripheral artery disease (STOP-PAD): Randomized, double-blind, placebo-controlled clinical trial. Vasc Med. 2019 Jun;24(3):200-207. doi: 10.1177/1358863X18817610. Epub 2019 Feb 21. PMID 30786835